CLINICAL TRIAL: NCT04839718
Title: Evaluating the Implementation and Outcomes of the Achieving Depression and Anxiety Patient Centered Treatment (ADAPT) Collaborative Care Program in A Large, Integrated Healthcare System: A Mixed Methods Observational Study Protocol
Brief Title: Evaluation of the Achieving Depression and Anxiety Patient Centered Treatment (ADAPT) Program
Acronym: ADAPT
Status: Withdrawn | Type: Observational
Why Stopped: Study redesigned to be a data-only cohort study and not a clinical trial prior to any patient recruitment activities.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 1421043
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients receiving referral to specialty mental healthcare
- ADAPT: ADAPT
  Interventions: Behavioral: ADAPT

INTERVENTIONS:
Behavioral: ADAPT — The Achieving Depression and Anxiety Patient Centered Treatment (ADAPT) Program is a novel collaborative psychiatric care model that is designed to unburden PCPs and psychiatrists, increase access to quality specialty mental healthcare for Kaiser Permanente members, and improve patient depression and anxiety treatment outcomes by utilizing technology-driven appointments. This program uses principles of collaborative care, including patient-centered care, population-based care, evidence-based care, measurement-based treatment to target, and accountable care.
  Groups: ADAPT

SUMMARY:
Depression and anxiety are increasingly common conditions for which primary care providers (PCPs) serve as the initial healthcare contact for most patients. Comorbid depression and anxiety result in higher costs, and treatment as usual, which is referrals to specialty psychiatric care, often contribute to delays in care. Collaborative psychiatric care is an evidence-based strategy to increase mental healthcare access while reducing costs. ADAPT is a novel collaborative care model. By using technology-driven appointments with providers, ADAPT increases access to mental healthcare, and reduces member wait times. This mixed methods study will assess implementation measures of the ADAPT program and the components of ADAPT related to patient mental health improvement compared to specialty mental health care. The hypothesis is that: ADAPT program will have good program reach and efficacy. We will examine program implementation and maintenance. Further, the study looks to uncover member and program characteristics that are associated with depression and anxiety remission and care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Adult Outcomes Questionnaire (AOQ) score between 10-30
* English-Speaking

Exclusion Criteria:

* High risk for suicide defined by answer to question 9 on PHQ-9 of 1 or more
* Diagnosis of bipolar disorder
* Diagnosis of a psychotic disorder
* Dementia diagnosis
* Active substance use disorder diagnosis
* Current hospice
* Current home-based palliative care
* Residing in a skilled nursing facility
* Residing in an assisted living facility
* Non-Kaiser Permanente Member
* Established psychiatric care outside of Kaiser Permanente

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kaiser Permanente Northern California adult members who screen positive for depression or anxiety in primary care and are referred to treatment.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient reach | through study completion, 2 years
  Examine and compare patients eligible and enrolled in ADAPT versus those eligible but not enrolled in ADAPT

SECONDARY OUTCOMES:
Member characteristics associated with depression remission | baseline, 3 and 6 months
  Clinical variables important to predicting intervention response: Patient demographics (age, sex, race/ethnicity, socioeconomic status), behavioral characteristics (exercise, sleep), and other individual characteristics (comorbidities, adverse childhood experiences, social supports, resilience).
Member characteristics associated with anxiety remission | baseline, 3 and 6 months
  Clinical variables important to predicting intervention response: Patient demographics (age, sex, race/ethnicity, socioeconomic status), behavioral characteristics (exercise, sleep), and other individual characteristics (comorbidities, adverse childhood experiences, social supports, resilience).
Efficacy: Patient therapy engagement | baseline, 3 and 6 months
  number of therapy contacts (individual, group and combined)
Efficacy: Patient medication provider engagement | baseline, 3 and 6 months
  number of clinical pharmacy contacts
Efficacy: Patient medication engagement | baseline, 3 and 6 months
  medication length of treatment
Efficacy: Patient psychiatry engagement | baseline, 3 and 6 months
  number of contact with psychiatrist
Efficacy: Patient time to care | baseline, 3 and 6 months
  average time from ADAPT referral to first appointment with therapist or pharmacist
Efficacy: Depression outcomes | baseline, 3 and 6 months
  Examine if patients enrolled in ADAPT demonstrate non-inferior depression outcomes defined by change in the patient health questionnaire (PHQ-9) score compared to treatment as usual.
Efficacy: Anxiety outcomes | baseline, 3 and 6 months
  Examine if patients enrolled in ADAPT demonstrate non-inferior anxiety outcomes defined by generalized anxiety disorder (GAD-2) score compared to treatment as usual.
Efficacy: Time to clinical improvement | baseline, 3 and 6 months
  Compare time to clinical improvement as defined by change in Adult Outcomes Questionnaire (AOQ score) from baseline to 3, and 6 months for members in ADAPT compared to treatment as usual.
Implementation: measurement-based care | through study completion, 2 years
  Examine provider use of measurement-based care
Implementation: Diagnosis | through study completion, 2 years
  Examine provider use of a specific depression or anxiety diagnosis
Maintenance: Measurement-based care | through study completion, 2 years
  Examine provider use of measurement-based care over time
Maintenance: Diagnosis | through study completion, 2 years
  Examine provider use of a specific depression or anxiety diagnosis over time

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn K Erickson-Ridout, MD PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No